CLINICAL TRIAL: NCT07231653
Title: Home Monitoring Study for Surgical Patients
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00146230
Record Dates: First submitted 2025-09-22; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Patient Monitoring; Postoperative Period
Keywords: Wellvii VitalDetect; Remote patient monitoring; Postoperative monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Home Monitoring - Surgical Patients
  Interventions: Device: Home-based Vital Sign Monitoring

INTERVENTIONS:
Device: Home-based Vital Sign Monitoring — Postoperative surgical patient will use the Wellvii VitalDetect, an FDA-cleared, non-invasive, handheld device for home-based monitoring of blood pressure, pulse rate, and temperature. After receiving training at discharge and recording baseline vital signs in clinic, participants will monitor their vital signs twice daily for two weeks using the device and a companion mobile app. Weekly clinic visits will collect corroborating data. The device does not requires calibration or maintenance and provides results in under 90 seconds. Usability and satisfaction will be assessed through questionnaires, and compliance will be monitored via app logs. Data will be automatically uploaded to a secure, de-identified database for analysis.

SUMMARY:
This clinical trial is designed to evaluate the accuracy, usability, and patient compliance of the Wellvii VitalDetect, an FDA-cleared (510(k) K231625), Class II medical device intended for non-invasive monitoring of vital signs including blood pressure, pulse rate, and temperature. The study will focus on comparing measurements obtained in a home environment using the device to those collected in a clinical setting, with the goal of validating the device's performance for real-world, at-home use.

The Wellvii VitalDetect is a portable, battery-operated, spot-check monitor that uses finger-based technology for most parameters and an infrared sensor for forehead-based, non-contact temperature readings. It is designed for use by adults (18 years or older) in a home environment and is not intended for continuous monitoring. In addition to the cleared vital signs, the device displays other wellness parameter for general health tracking. A smartphone application supports the user experience by delivering usage instructions and data display.

The study will assess:

* Measurement accuracy compared to standard clinical instruments
* Patient ease-of-use and engagement with the device
* Adherence to regular self-monitoring schedules
* Overall user satisfaction and confidence I home-based monitoring

This research will contribute to the growing body of evidence supporting remote patient monitoring solutions and aims to advance the adoption of decentralized technology-enabled healthcare delivery.

The study aligns with Wellvii Inc.'s mission to transform healthcare delivery by enabling continuous, connected health monitoring from the home. The ultimate goal is to empower patients and healthcare providers with real-time, clinically actionable health at a that can lead to earlier intervention, improved outcomes, and reduced system burden.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients requiring routine postoperative monitoring in the absence of any acute illness following surgery.
* Able to use a smartphone or tablet for the monitoring system.

Exclusion Criteria:

* Severe cognitive impairment or conditions that may interfere with the use of home monitoring devices.
* Currently participation in other clinical trials involving vital sign monitoring.
* Unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical procedures, including day surgery procedures and those procedures requiring a hospital stay
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Home-Based Vital Sign Monitoring Compared to Standard Clinical Measurements | For a two-week period (twice daily) following their discharge from hospital.
  This outcome measures the accuracy of vital sign readings (temperature, blood pressure, and heart rate) collected at home using the Wellvii VitalDetect™ compared to standard clinical equipment readings taken during weekly hospital visits. Accuracy will be evaluated using paired t-tests to compare mean differences between home and clinical measurements.

SECONDARY OUTCOMES:
Patient Compliance with Home Monitoring Protocol | At one and two weeks post-hospital discharge
  This outcome assess participant compliance with the home monitoring protocol, defined as the percentage of days during the two-week study period in which complete vital sign measurements are successfully recorded using the device and app.

OTHER OUTCOMES:
Patient satisfaction with Home Monitoring Protocol | At the one-week and two-week clinic visits
  Satisfaction will be assessed using a Likert-scale questionnaire. The questionnaire evaluates overall satisfaction with the device.

CONTACTS AND LOCATIONS:
Overall Officials: Todd McMullen, MD, Principal Investigator — Mackenzie Health Science Centre, University of Alberta
Locations (1):
- Mackenzie Health Science Centre, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No